CLINICAL TRIAL: NCT01652365
Title: Evaluation of the Feasibility and Impact of Introducing Malaria Rapid Diagnostic Tests in the Retail Sector: A Randomized Controlled Trial in Eastern Uganda
Brief Title: Feasibility and Impact of Malaria Rapid Diagnostic Tests in the African Retail Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Clinton Health Access Initiative, Nigeria (Other); Innovations for Poverty Action-Uganda (Unknown); Uganda Health Marketing Group (Unknown)
Responsible Party: Principal Investigator, Jessica Cohen, Assistant Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 19371-106; HS805 (Other: Uganda National Council for Science and Technology)
Record Dates: First submitted 2012-07-24; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Malaria
Keywords: Malaria Diagnosis; Rapid Diagnostic Tests; RDTs; Private Sector; Retail Sector; Drug Shops
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDT Training and Subsidy Offered (Experimental): Licensed drug shops within villages selected randomly to be in this arm will be invited to training on RDTs and offered access to subsidized RDTs available for purchase at a local wholesale pharmacy in Mbale, Uganda.
  Interventions: Behavioral: RDT Training and Subsidy Offered
- Information/Education Campaign (Experimental): Community meetings describing RDTs and encouraging community members to be diagnosed prior to taking malaria treatment will be held in villages randomly assigned to this treatment arm.
  Interventions: Behavioral: Information/Education Campaign
- RDT Training/Subsidy + Information/Education Campaign (Experimental): Includes both the training and subsidy component and the information/education campaign component.
  Interventions: Behavioral: RDT Training and Subsidy Offered; Behavioral: Information/Education Campaign
- Control (No Intervention)

INTERVENTIONS:
Behavioral: RDT Training and Subsidy Offered
  Arms: RDT Training and Subsidy Offered; RDT Training/Subsidy + Information/Education Campaign
Behavioral: Information/Education Campaign
  Arms: Information/Education Campaign; RDT Training/Subsidy + Information/Education Campaign

SUMMARY:
The purpose of this study is to assess the feasibility and impact of introducing subsidized malaria rapid diagnostic tests (RDTs) into retail sector drug shops in Uganda. This is a randomized controlled trial at the village level, taking place in 6 districts in Eastern Uganda. Licensed drug shops in selected villages were trained in proper RDT storage, administration, interpretation and disposal and were given access to subsidized RDTs for sale. This study explores whether drug shop owners--when given access to training and subsidized RDTs--will choose to promote and sell RDTs to customers and, if so, at what volume and what price. The investigators also explore whether shops will safely store, administer, interpret and dispose of RDTs and to what extent they will use RDT results to guide treatment recommendations. Finally, the study explores whether making RDTs available for sale in local drug shops has a community level impact on diagnostic testing and appropriate treatment for malaria.

ELIGIBILITY:
Inclusion Criteria:

Drug Shops:

* Licensed and registered as a Drug Shop with the Ugandan National Drug Authority

Households:

* Live in the village of participating drug shop
* Female household head is 18 or over

Exclusion Criteria:

Drug Shops:

* Drug Shop not registered with Ugandan National Drug Authority
* Female household head is under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Fraction of Illnesses Diagnosed for Malaria | Up To One Year
  Comparison of the rate of malaria diagnosis in treatment vs. control. Comparison will be at the village level and at the shop level. Denominator will be: all illnesses, febrile illnesses only or suspected malaria episodes only.

SECONDARY OUTCOMES:
Mean RDT Price Charged by Shops | Up to One Year
Mean RDTs Purchased by Shops from Wholesaler | Up To One Year
Fraction of Monitoring Checklist Items Performed Correctly by Shops | Up To One Year
Fraction of Illnesses for which an Antimalarial/ACT/Antibiotic is Taken | Up To One Year
  * Comparison of rate of antimalarial taking for illnesses in treatment vs. control
  * Comparison of rate of ACT taking for illnesses in treatment vs. control
  * Comparison of rate of antibiotic taking for illnesses in treatment vs. control

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cohen, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Gunther Fink, PhD, Principal Investigator — Harvard School of Public Health (HSPH); William Dickens, PhD, Principal Investigator — Northeastern University
Locations (2):
- Uganda (2):
  - Clinton Health Access Initiative, Kampala
  - Innovations for Poverty Action-Uganda, Kampala

REFERENCES:
- See also: Project Description — http://www.poverty-action.org/project/0508
- See also: G Fink (PI) website — http://www.hsph.harvard.edu/faculty/gunther-fink/